CLINICAL TRIAL: NCT05293704
Title: An Open Study on the Preventive Effect of Early Mizoribine Conversion on BKV Nephropathy in Renal Transplant Recipients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BLDN-LEES-2022-3
Record Dates: First submitted 2022-03-12; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Kidney Transplant Recipients; BK Virus
MeSH Terms: interventions — mizoribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Mizoribine — Orally administered at 3-4 mg/kg/d, once every 12 hours; When body weight ≤50 kg, each dose of 75 mg; Weight & gt At 50 kg, the dosage was 100 mg each time.

SUMMARY:
This study is divided into two parts: ① Part I was a retrospective observational study. Kidney transplant recipients infected with BK virus (BKV) in the First Affiliated Hospital of Sun Yat-sen University from 2015 to 2021 were retrospectively collected and divided into case group and control group whether to convert MPA drug to mizoribine. ② The second part was a prospective, open and interventional clinical trial. Thirty patients with positive urinary BK virus after kidney transplantation using Mycophenolic acid (MPA) were enrolled in the First Affiliated Hospital of Sun Yat-sen University. All patients who met the inclusion criteria were treated with mizoribine to place MPA (Mycophenolate or mycophenolate sodium enteric coated tablets) for 12 months as directed. At the baseline of follow-up (before enrollment) and at each follow-up point, clinical indicators of patients were recorded, and renal biopsy was performed to evaluate the occurrence of BKV nephropathy in patients with persistent elevated BK viruria or persistent BK viremia after conversion and patients with BK viruria after 12 months, and to judge the progress after early activation of BKV and the safety of mizoribine.

DETAILED DESCRIPTION:
This study is divided into two parts: ① Part I was a retrospective observational study. Kidney transplant recipients infected with BK virus (BKV) in the First Affiliated Hospital of Sun Yat-sen University from 2015 to 2021 were retrospectively collected and divided into case group and control group whether to convert MPA drug to mizoribine. The basic data of the two groups, the concentration of mizoribine, the clinical benefit after conversion and the outcome of BKV infection were analyzed, and the clinical improvement rate and preliminary safety of mizoribine conversion on BKV infection were determined. ② The second part was a prospective, open and interventional clinical trial. Thirty patients with positive urinary BK virus after kidney transplantation using Mycophenolic acid (MPA) were enrolled in the First Affiliated Hospital of Sun Yat-sen University. The patients and their families voluntarily participated in the experiment and signed the Informed Consent on the premise of fully understanding the treatment plan. The treatment was approved by the hospital ethics Committee. All patients who met the inclusion criteria were treated with MPA (Mycophenolate or mycophenolate sodium enteric coated tablets) replaced with mizoribine for 12 months. At the baseline of follow-up (before enrollment) and at each follow-up point, clinical indicators of patients were recorded, and renal biopsy was performed to evaluate the occurrence of BKV nephropathy in patients with persistent elevated BK viruria or persistent BK viremia after conversion and patients with BK viruria after 12 months, and to judge the progress after early activation of BKV and the safety of mizoribine.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients;
* Postoperative maintenance therapy with glucocorticoid + tacrolimus +MPA;
* Urinary BKV-DNA load ≥10^7/L;
* No gender limitation for recipients > 18 years of age;
* Voluntarily sign written informed consent.

Exclusion Criteria:

* Multiple organ transplantation;
* Acute rejection occurred within 1 week before enrollment;
* Recipients with signs of active infection;
* Recipients with white blood cell count below 3,000 /cubic metre;
* Women who are pregnant, breast-feeding, or unwilling to use appropriate contraceptive methods during the study period;
* Patients with serious gastrointestinal diseases and active peptic ulcer disease;
* Suffering from any mental illness;
* Patients with severe heart disease and abnormal cardiac function;
* Subjects with known allergy to the test drug;
* Other competent physicians judged that the recipients were not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who had BKV-related nephropathy occurred | 12 month
  During the follow-up, patients with urinary BKV-DNA increase of more than 10 times for 3 consecutive months after dressing change, or viremia (serum BKV-DNA load ≥10^4/ mL) for 3 consecutive months after dressing change, as well as patients with urinary BKV positive 12 months after dressing change, were evaluated by renal biopsy pathology. The number of Participants who had BKV-related nephropathy occurred will be counted.（BKV stands for BK polyoma virus）

SECONDARY OUTCOMES:
Number of Participants in who Serum and urine BK viral load were cleared | 12 month
  During the observation period, the presence of serum BKV and the corresponding BKV-DNA load of the subjects were recorded to determine the incidence and outcome of BKV.
Number of Participants with Acute rejection | 12 month
  Diagnosis of acute rejection: including clinical diagnosis and pathological diagnosis. If the serum creatinine increased by more than 20% within 72 hours, acute rejection was suspected, and ultrasound examination of the transplanted kidney was performed, and biopsy of the transplanted kidney was performed if necessary. Acute rejection (BPAR) confirmed by biopsy needs to be diagnosed by a pathologist according to the classification criteria (1997 edition and subsequently updated). If not confirmed by biopsy, acute rejection should be diagnosed based on the exclusion of other causes of elevated creatinine.
Number of Participants with Renal graft loss | 12 month
  During the study, renal function was recorded, the survival of transplanted kidneys was counted and the survival rate of transplanted kidneys was calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided